CLINICAL TRIAL: NCT00838448
Title: Interactions Between Physical Activity and Cannabis Use in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Maciej Buchowski, Research Professor, Vanderbilt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 081302
Record Dates: First submitted 2009-01-23; First posted 2009-02-06 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Cannabis Dependence
Keywords: exercise; cannabis use; visual cues
MeSH Terms: conditions — Marijuana Abuse; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cannabis users (Experimental): Cannabis users
  Interventions: Behavioral: Exercise
- Cannabis no-users (Experimental): Cannabis no-users
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise performed on a treadmill for 20-30 minutes

SUMMARY:
In this study the investigators will explore the relationship between physical activity and cannabis use. The investigators will compare regional brain activation detected by imaging technique(fRMI) before and after exercise in cannabis users and compare results with results from controls. The investigators hypothesize that the regional brain activation in response to visual cues (pictures related to cannabis use and food) will be different in cannabis users than in controls and that exercise will significantly alter brain responses to the cues.

DETAILED DESCRIPTION:
It is unknown how the response of cannabis users might compare to those of non-users in response to similar dose of physical activity. We will therefore compare brain activation during craving to cannabis, a natural reward (food) and a neutral scene (nature images). The food cues will allow us to determine if effects of exercise on brain activation and craving generalize to two different reward conditions and the nature scenes provide a neutral, no rewarding control. In addition to the analysis of predetermined regions of interest, whole-brain exploratory analyses will also be conducted to examine for additional brain regions showing associations between various conditions of interest and regional brain activation.

Specific Aims

1. To explore methodological factors involved in finding the relationship between PA and cannabis use.

1. to examine the effects of cannabis and food cues on brain activation and craving in cannabis users and nonusers
2. to examine the effects of vigorous exercise on brain activation and craving in response to cannabis and food cues.

Our working hypothesis is that the regional brain activation in response to drug cues will be different in cannabis users than in controls and that exercise will significantly alter brain responses to these cues in both groups. Our secondary hypothesis is that exercise will tend to normalize the abnormal brain activation observed in cannabis users.

Our expectation is that exercise will alter cue-responding in terms of brain activation or craving. It is possible that exercise may be a useful treatment in cannabis dependence. Future studies may examine this specific relationship.

There are no reports available exploring the relationship between physical activity and cannabis use.

Current data suggest that there are convergent findings regarding the chronic and acute effects of cannabis on brain activity

ELIGIBILITY:
Inclusion Criteria:

* Cases and Controls must:

  * Be able to understand the study and provide written informed consent.
  * Be male or female 18 -35 years of age.
  * Be in generally good health
  * If female of childbearing potential, have a negative serum pregnancy test on study day

Cases must:

* Meet criteria for cannabis dependence as primary diagnosis as determined by the Substance Abuse module of SCID (Structured Clinical Interview for DSM-IV).
* Not currently seeking treatment for cannabis dependence.
* Have a positive urine drug test for cannabis on the study day
* Avoid alcohol and other recreational drug use (except cannabis and/or nicotine) for 48 h before testing.

Exclusion Criteria:

* Cases and Controls must not:

  * Be pregnant or lactating
  * Have implanted electrical medical device (e.g. pacemaker, vagal nerve stimulator)
  * Have non-secure metallic foreign bodies
  * Have met criteria for another axis 1 diagnosis in the past 6 months
  * Receive psychotropically active or vasoactive medications (within 6 weeks of screen day)
  * Have chronic medical illness
  * Have epilepsy
  * Have a history of head injury that required hospitalization
  * Have claustrophobia
  * Have orthopedic or other problems precluding them from performing exercise protocol
  * Have body mass index (BMI) less than 19 kg/m2
  * Weighing more than 275 pounds (MRI table limit)

Cases must not:

* Have current dependence, as determined by the SCID, on any psychoactive substance other than nicotine and/or cannabinoid
* Have any serious medical or psychiatric illnesses and/or clinically significant symptoms, which in the judgment of the PI or his/her designee would make them unsafe, or would make compliance with the study protocol difficult or put the study staff at undue risk

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Craving for cannabis | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Maciej S Buchowski, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Charboneau EJ, Dietrich MS, Park S, Cao A, Watkins TJ, Blackford JU, Benningfield MM, Martin PR, Buchowski MS, Cowan RL. Cannabis cue-induced brain activation correlates with drug craving in limbic and visual salience regions: preliminary results. Psychiatry Res. 2013 Nov 30;214(2):122-31. doi: 10.1016/j.pscychresns.2013.06.005. Epub 2013 Sep 12. PMID 24035535
- [Derived] Buchowski MS, Meade NN, Charboneau E, Park S, Dietrich MS, Cowan RL, Martin PR. Aerobic exercise training reduces cannabis craving and use in non-treatment seeking cannabis-dependent adults. PLoS One. 2011 Mar 8;6(3):e17465. doi: 10.1371/journal.pone.0017465. PMID 21408154